CLINICAL TRIAL: NCT01611597
Title: Continuous Measurement of the Activity for Clinical Evaluation at Home, for Non-ambulant Neuromuscular Patients
Acronym: Pre-Acti
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut de Myologie, France (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: Pre-Acti
Record Dates: First submitted 2012-05-30; First posted 2012-06-05 (Estimated); Last update posted 2013-04-19 (Estimated); Status verified 2013-04

CONDITIONS: Neuromuscular Disease
Keywords: accelerometry; neuromuscular disease
MeSH Terms: conditions — Neuromuscular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Different standardized tasks with an accelerometer device — Patients will perform tests like hand grip (MyoGrip), pinch (MyoPinch), Moviplate, box and block test of hand function, Minnesota Manual Dexterity Test. The tests will be performed with the accelerometer device worn on the wrist.
  Other Names: MyoGrip; MyoPinch; Moviplate

SUMMARY:
Validation of a measure specifically suitable to evaluate the residual function of upper limbs of non-ambulant neuromuscular patients, especially with Duchenne muscular dystrophy and spinal muscular atrophy.

This approach is of fundamental importance for clinical monitoring and preparing the future therapeutic trials.

DETAILED DESCRIPTION:
The main objective is the continuous measurement of muscle activity in a standardized setting and in the non ambulatory patient's natural environment. This measure uses an innovative technology based on accelerometer and magneto-inertial sensors. The system is intended to measure the physical activity of patients from the extraction of data recorded by the sensors in the three space axes.

The non ambulatory patients will be included and evaluated at baseline and 14 days later. The patients wear the accelerometer device during some standard evaluations and also at home continuously for 14 days.

With this protocol the investigators want to try to find the best variable that characterizes the movement of the upper limbs of non-ambulant neuromuscular patients.

The aim of Pre-Acti is to propose a primary outcome measure that may be used in clinical monitoring of patients.

ELIGIBILITY:
Inclusion Criteria:

* age over 10 years
* neuromuscular disease documented by genetic testing or by muscle biopsy
* not able to walk 10 meters without support
* capable of sitting upright in a wheelchair for at least 3 hours
* subject affiliated to a social security system
* subject who signed an informed consent

Exclusion Criteria:

* severe intellectual impairment limiting the comprehension of the demanded tasks
* acute neurologic, inflammatory, infectious, endocrine, orthopedic disease in the month preceding the inclusion
* surgery scheduled within 3 weeks after enrollment
* surgery at upper limbs in the three months preceding the inclusion
* pregnant or nursing women

Ages: 10 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2012-01; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Physical activity variables of upper limbs movement at home | each day for 14 days
  A watch containing and inertial system will be worn by non-ambulant patients with neuromuscular diseases at home for 14 days. Physical activity variables will be deduced from these measurements.

SECONDARY OUTCOMES:
Physical activity variables of upper limbs movement in standardized setting | at baseline
  A watch containing and inertial system will be worn by non-ambulant patients with neuromuscular diseases during standardized tasks. Physical activity variables will be deduced from these measurements.
Physical activity variables of upper limbs movement in standardized setting | 14 days after baseline
  A watch containing and inertial system will be worn by non-ambulant patients with neuromuscular diseases during standardized tasks. Physical activity variables will be deduced from these measurements.

CONTACTS AND LOCATIONS:
Overall Officials: Laurent Servais, MD, PhD, Principal Investigator — institut de myologie
Locations (1):
- Institut de Myologie - GH Pitié Salpétrière, Paris, France

REFERENCES:
- [Derived] Le Moing AG, Seferian AM, Moraux A, Annoussamy M, Dorveaux E, Gasnier E, Hogrel JY, Voit T, Vissiere D, Servais L. A Movement Monitor Based on Magneto-Inertial Sensors for Non-Ambulant Patients with Duchenne Muscular Dystrophy: A Pilot Study in Controlled Environment. PLoS One. 2016 Jun 7;11(6):e0156696. doi: 10.1371/journal.pone.0156696. eCollection 2016. PMID 27271157